CLINICAL TRIAL: NCT01385787
Title: The Role of Minimal Residual Disease Testing Before and After Hematopoietic Cell Transplantation for Pediatric Acute Myeloid Leukemia
Brief Title: MRD Testing Before and After Hematopoietic Cell Transplantation for Pediatric Acute Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: Center for International Blood and Marrow Transplant Research (Network)
Collaborators: Pediatric Blood and Marrow Transplant Consortium (Other); St. Baldrick's Foundation (Other); Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 09-MRD
Record Dates: First submitted 2011-06-28; First posted 2011-06-30 (Estimated); Last update posted 2017-09-07 (Actual); Status verified 2017-09

CONDITIONS: Acute Myeloid Leukemia
Keywords: Pediatric (ages 0-21 years); myeloablative HCT; PBMTC sites
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is a non-therapeutic study. Pediatric AML patients undergoing HCT with a myeloablative preparative regimen may be enrolled. Subjects can be enrolled 10-40 days prior to HCT. Three samples for MRD (measured by WT1 PCR and flow cytometry) will be collected from peripheral blood and bone marrow: 1) pre-HCT (<3 weeks prior to starting the preparative regimen), 2) day 42 +/- 14 days post HCT (early post-engraftment), and 3) day 100 (+/-20 days) post HCT. For two years after transplant, the subject's follow-up data will be collected using the Research Level Forms in the CIBMTR Forms Net internet data entry system. The main objective is to determine whether there is any association between level of pre-transplant and post-transplant bone marrow MRD using WT1 and flow cytometry with 2-year event-free-survival, and to estimate the strength of that association in terms of the predictive accuracy of MRD. The investigators hypothesize that measurable MRD at either time point will be associated with decreased 2-year event-free survival.

DETAILED DESCRIPTION:
This is a prospective, non-therapeutic study, assessing the significance of minimal residual disease (MRD) at three different time points in relation to allogeneic HCT for pediatric AML. The study is a collaboration between the Pediatric Blood and Marrow Transplant Consortium (PBMTC) and the Resource for Clinical Investigations in Blood and Marrow Transplantation (RCI-BMT) of the Center for International Blood and Marrow Transplant Research (CIBMTR). The study will enroll pediatric AML patients who undergo myeloablative HCT at PBMTC sites. The eligibility criteria for this non-therapeutic study mirror widely accepted criteria for allogeneic HCT in pediatric AML.

The study tests the hypothesis that assessment of pre-transplant and post-transplant MRD predicts 2-year outcomes following transplant. Two MRD methodologies are being studied: flow cytometry and WT1 PCR. The secondary hypothesis is that combining these 2 methodologies will improve the accuracy in predicting 2-year outcomes following transplant.

It is well established that the level of minimal residual disease (MRD) during chemotherapy is a strong predictor of relapse in children with acute lymphoblastic leukemia (ALL) [33, 34]. Within this population, MRD levels have the potential to predict those patients who will respond well to standard therapy, thus allowing clinicians to tailor therapy and minimize toxicity while ensuring maximal cure rates [10]. MRD levels before allogeneic hematopoietic stem cell transplantation (HCT) also predict the risk of relapse post-HCT [25], leading to the clinical practice of reducing MRD levels as much as possible before transplant. By contrast, in children with acute myeloid leukemia (AML), the prognostic value of MRD levels prior to HCT remains unclear.

Our long-term objective is to improve the cure rate for children with AML. The investigators hypothesize that MRD levels before HCT will provide a powerful tool to select the best candidates for transplant, guide decision making in stem cell source and preparative therapy, and optimize the timing of the transplant. Measurements of MRD post-HCT will allow informed decisions about withdrawal of immunosuppressive therapy, administration of donor lymphocyte infusions, or alternative targeted therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Subject or legal guardian to understand and voluntarily sign an informed consent.
2. Age 0-21 at time of transplant.
3. Karnofsky score ≥ 70% (age ≥ 16 years old), or Lansky score ≥ 70% (age<16 years old).
4. Patients with adequate physical function as measured by:

   * Cardiac: Left ventricular ejection fraction at rest must be > 40%, or shortening fraction > 26%
   * Hepatic: Bilirubin ≤ 2.5 mg/dL; and ALT, AST and Alkaline Phosphatase≤ 5 x ULN
   * Renal: Serum creatinine within normal range for age, or if serum creatinine outside normal range for age, then renal function (creatinine clearance or GFR) > 70 mL/min/1.73 m2.
   * Pulmonary: DLCO, FEV1, FVC (diffusion capacity) > 50% of predicted (corrected for hemoglobin); if unable to perform pulmonary function tests, then O2 saturation > 92% in room air.
5. Acute myelogenous leukemia (AML) at the following stages:

   * High risk first complete remission (CR1), defined as:

     * Having preceding myelodysplasia (MDS) -or-
     * Diagnostic high risk karyotypes: del (5q) -5, -7, abn (3q), t (6;9), abnormalities of 12, t (9:22), complex karyotype (≥3 abnormalities), the presence of a high FLT3 ITD-AR (> 0.4) -or-
     * Having >15% bone marrow blasts after 1st cycle and/or >5% after 2nd cycle before achieving CR -and-
     * <5% blasts in the bone marrow, with peripheral ANC>500
   * Intermediate risk first complete remission (CR1), defined as:

     * Diagnostic karyotypes that are neither high-risk (as defined above) nor low risk (inv(16)/t(16:16); t(8;21); t(15;17)). Included are cases where cytogenetics could not be performed. -and-
     * <5% blasts in the bone marrow, with peripheral ANC>500
   * High risk based upon COG AAML 1031 criteria:

     * High allelic ratio FLT3/ITD+, monosomy 7, del(5q) with any MRD status or standard risk cytogenetics with positive MRD at end of Induction I.
     * <5% blasts in the bone marrow, with peripheral ANC>500
   * Second or greater CR

     * <5% blasts in the bone marrow, with peripheral ANC>500
   * Therapy-related AML at any stage

     * Prior malignancy in remission for >12 months.
     * <5% blasts in the bone marrow, with peripheral ANC>500
6. Myeloablative preparative regimen, defined as a regimen including one of the following as a backbone agent*:

   * Busulfan ≥ 9mg/kg total dose (IV or PO). PK-based dosing is allowed, if intent is myeloablative dosing OR
   * Total Body Irradiation≥1200cGy fractionated OR
   * Treosulfan ≥ 42g/m2 total dose IV *Regimens may include secondary agents such as, but not limited to Ara-C, Fludarabine, VP-16. Regimens that combine Busulfan and TBI or treosulfan and TBI are allowed as long as the Busulfan or treosulfan meets or exceeds the dose listed and the TBI is below the dose listed.
7. Graft source:

   * HLA-identical sibling PBSC, BM, or cord blood
   * Adult related or unrelated donor PBSC or BM matched at the allelic level for HLA-A, HLA-B, HLA-C, and HLA-DRB1 with no greater than a single antigen mismatch.
   * One or two unrelated cord blood units:

     * HLA≥4:6 at the low resolution level for HLA-A, HLA-B, at high resolution level at HLA-DRB1 for one or both units.
     * If one unit, must have TNC≥2.5x107/kg; if two units, combination of the two must have TNC≥2.5x107/kg

Exclusion Criteria:

1. Women who are pregnant (positive HCG) or breastfeeding.
2. Evidence of HIV infection or HIV positive serology.
3. Positive viral load (PCR) for Hepatitis B or C (negative serology, surface antigen, and core antibody may substitute for PCR).
4. Current uncontrolled bacterial, viral or fungal infection (currently taking medication and progression of clinical symptoms).
5. Autologous transplant < 12 months prior to enrollment.
6. Prior allogeneic hematopoietic stem cell transplant.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participating institutions (transplant centers)
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Two-year Event Free Survival (EFS) | 2 years post-HCT
  Event-free survival is defined as the time from HCT to relapse, death, initiation of post-HCT therapy to treat AML relapse, loss to follow up or end of study whichever comes first.

SECONDARY OUTCOMES:
Two-year overall survival (OS) | 2 years post-HCT
  Overall survival is the time from HCT to death from any cause, loss to follow up or end of study, whichever comes first.
Disease relapse at 2 years | 2 years post-HCT
  Relapse includes morphologic reappearance of leukemia or treatment for impending relapse. Death in remission is a competing risk. Relapse is defined as in 3.1. Cytogenetic or molecular relapse with <5% leukemic blasts in the bone marrow does not constitute a relapse unless unplanned AML-directed therapy is administered.
Occurrence of acute grade II-IV and grade III-IV GVHD by 200 days post-HCT | 200 days post-HCT
  Any skin, gastrointestinal or liver abnormalities fulfilling the consensus criteria [36] of grades II-IV or grades III-IV acute GVHD are considered events. Death and second transplants are competing risks, and patients alive without acute GVHD will be censored at the time of last follow-up.
Occurrence of chronic GVHD at 2 years post-HCT | 2 years post-HCT
  Occurrence of any symptoms in any organ system fulfilling the CIBMTR criteria of limited or extensive chronic GVHD. Death and the second transplant are competing risks, and patients alive without chronic GVHD will be censored at time of last follow-up.
Time to neutrophil engraftment | 42 days post-HCT
  1st consecutive day of a sustained ANC ≥ 500/ μL for 3 consecutive days. Death without engraftment and second transplants are considered competing risks.
Time to platelet engraftment | 42 days post-HCT
  1st day of platelet count ≥20,000/μL that persists ≥7 days, without transfusion. Death without engraftment and second transplants are considered competing risks.
Veno-occlusive Disease | 2 years post-HCT
  Cumulative incidence of veno-occlusive disease (VOD)/sinusoidal obstruction syndrome (SOS), with median maximum bilirubin for subjects diagnosed with VOD/SOS. Subjects classified as having had VOD/SOS must meet the Jones Criteria, defined as: bilirubin>2mg/dL and at least 2 of the following signs: a) hepatomegaly and/or right upper quadrant pain, and b) >5% weight gain.
Chimerism | 100 days post-HCT
  Whole blood chimerism and T-cell chimerism will be classified according to full (>95%), mixed (5-95%), or none (<5%) at 100 days.

CONTACTS AND LOCATIONS:
Overall Officials: David A. Jacobsohn, MD, ScM, Principal Investigator — Children's National Research Institute
Locations (38):
- United States (34):
  - The Children's Hospital of Alabama, University of Alabama at Birmingham, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Loma Linda University, Loma Linda, California
  - University of California San Francisco, San Francisco, California
  - The Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Miami Children's Hospital, Miami, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Riley Hospital for Children/Indiana University, Indianapolis, Indiana
  - University of Louisville, Louisville, Kentucky
  - Johns Hopkins, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Washington University, St. Louis Children's Hospital, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Mount Sinai School of Medicine, New York, New York
  - Columbia University - The Morgan Stanley Children's Hospital of New York, New York, New York
  - New York Medical College, Valhalla, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - University Hospitals of Cleveland Case Medical Ctr, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health & Sciences University - Doerbecher Children's, Portland, Oregon
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Methodist Children's Hospital of South Texas/Texas Institute of Medicine and Surgery, San Antonio, Texas
  - University of Utah - Primary Children's Medical Center, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Canada (4):
  - Alberta Children's Hospital, Calgary, Alberta
  - Children's & Women's Health Centre of British Columbia, Vancouver, British Columbia
  - The Montreal Children's Hospital, Montreal, Quebec
  - Hopital Ste. Justine, Montreal, Quebec